CLINICAL TRIAL: NCT00108290
Title: Chemohormone Therapy Prior to Prostatectomy in High Risk Prostate Cancer
Brief Title: Chemotherapy, Hormone Therapy, and Surgery to Remove the Prostate Gland in Patients With High Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-003-02F
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; chemotherapy; hormone therapy; surgery; PSA; Gleason score
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Drug Therapy

INTERVENTIONS:
Drug: Chemotherapy

SUMMARY:
In men with prostate cancer who do not have evidence of spread to bone or other sites on computed axial tomography (CAT) scan/bone scan but are still at significant risk of failing treatment with surgery or radiation alone, a combination of chemotherapy and hormone therapy is being given for 6 months followed by surgery to remove the prostate.

ELIGIBILITY:
Inclusion Criteria:

* High risk prostate cancer without evidence of bone metastasis.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States